CLINICAL TRIAL: NCT02088710
Title: Clinical Cohort of Individual Expectations, Side Effects, Quality of Life and Adherence in Postoperative Women With Estrogen Receptor Positive Breast Cancer During Endocrine Therapy
Brief Title: Expectations and Side Effects of Endocrine Therapy in Women With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Yvonne Nestoriuc, PhD., Prof. Dr., Philipps University Marburg
Other Study IDs: BB-2011
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Female Breast Cancer
Keywords: Patients´ Expectations; Breast Cancer; Adjuvant Endocrine Treatment; Nocebo; Psycho-oncology; Satisfaction with information
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Enhanced information about endocrine therapy — Enhanced information about endocrine therapy, extending clinical routine information

SUMMARY:
The purpose of this study is to evaluate the role of patients' response expectations for nocebo side effects, quality of life and adherence during adjuvant endocrine treatment (AET). Furthermore, this study analyses the effects of a structured treatment information on patients' satisfaction with information, response expectations, knowledge and adherence.

DETAILED DESCRIPTION:
The majority of breast cancer patients discontinues today's standard adjuvant treatment (endocrine therapy) due to side effects and reduced quality of life. Thereby, most side effects are unspecific, suggesting a role of psychological factors as patients´ expectations (nocebo effects). Moreover, patients are not informed sufficiently about their treatment.

Using a longitudinal design, the nature and onset of adverse side effects and their association to treatment related expectations are investigated. Postoperative patients with hormone receptor-positive breast cancer are assessed before the start of adjuvant treatment. All patients receive standardized, additional information about endocrine therapy. Expectations about side effects, knowledge and satisfaction with the enhanced information are assessed before and after informing patients. Side effects, quality of life and adherence are measured three months, two and five years after start of medication intake.

It will be analyzed if patients' response expectations predict side effects and quality of life during medication intake to provide insights into pathways of clinical nocebo effects. Further, this study examines the effects of a structured treatment information on patients' satisfaction with information, response expectations, knowledge and adherence. The study findings promise significant advances in the clinical nocebo research with strong implications for clinical and research practice.

ELIGIBILITY:
Inclusion Criteria:

* Post surgery women with estrogen receptor positive breast cancer scheduled to start first-line adjuvant endocrine therapy with Tamoxifen (+/- GnRH) or a third generation Aromatase inhibitor at the Breast Cancer Centre
* Sufficient knowledge of German language and ability to give informed consent
* Age of 18 and more

Exclusion Criteria:

* Presence of a serious comorbid psychiatric condition (schizophrenia or addiction, severe depression or anxiety)
* Presence of a life threatening comorbid medical condition

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Side Effects | up to 5 years
  General Assessment of Side Effects (GASE)

SECONDARY OUTCOMES:
Quality of Life | up to 5 years
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) with breast module (QLQ-BR23)
Adherence | up to 5 years
  Medication Adherence Report Scale (MARS-D); Adherence with endocrine treatment; reasons for non-adherence
Knowledge | up to 5 years
  Patients' knowledge of hormone receptor status of their tumor
Satisfaction with Information | Baseline
  Satisfaction with Information about Medicines Scale, (SIMS-D)
Expectations | Baseline
  General Assessment of Side Effects Scale - Expectations Module
Coping with Side Effects | Follow-up (3 months, 2 years, 5 years)
  General Assessment of Side Effects Scale -Coping Module

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nestoriuc, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Winfried Rief, Prof. Dr., Study Chair — Philipps University Marburg
Locations (1):
- Philipps University Marburg Medical Center, Marburg, Hesse, Germany

REFERENCES:
- [Derived] Pan Y, Heisig SR, von Blanckenburg P, Albert US, Hadji P, Rief W, Nestoriuc Y. Facilitating adherence to endocrine therapy in breast cancer: stability and predictive power of treatment expectations in a 2-year prospective study. Breast Cancer Res Treat. 2018 Apr;168(3):667-677. doi: 10.1007/s10549-017-4637-2. Epub 2018 Jan 12. PMID 29330625
- [Derived] Nestoriuc Y, von Blanckenburg P, Schuricht F, Barsky AJ, Hadji P, Albert US, Rief W. Is it best to expect the worst? Influence of patients' side-effect expectations on endocrine treatment outcome in a 2-year prospective clinical cohort study. Ann Oncol. 2016 Oct;27(10):1909-15. doi: 10.1093/annonc/mdw266. Epub 2016 Aug 22. PMID 27551051
- See also: Homepage of the research unit (FOR 1328): Expectation and conditioning as basic processes of the placebo and nocebo response: From neurobiology to clinical applications — http://www.placeboforschung.de/